CLINICAL TRIAL: NCT02652429
Title: An Open-Label Long-Term Safety Study of Inhaled Nitric Oxide (iNO) for PAH for Subjects in the PULSE-PAH-006 and PULSE-PAH-004 Studies Who Continue to Need iNO Therapy
Brief Title: Long-Term Extension Study of Inhaled Nitric Oxide (iNO) for PAH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bellerophon Pulse Technologies (Industry)
Responsible Party: Sponsor
Organization: Bellerophon (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PULSE-PAH-006
Record Dates: First submitted 2015-12-17; First posted 2016-01-11 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2022-02

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH; Pulmonary Arterial Hypertension; Inhaled Nitric Oxide; iNO
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Intervention Model Description: Open Label Extension
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Inhaled Nitric Oxide (iNO) (Experimental): Pulsed iNO 75 mcg/kg IBW/hour
  Interventions: Drug: Inhaled Nitric Oxide

INTERVENTIONS:
Drug: Inhaled Nitric Oxide
  Other Names: iNO

SUMMARY:
An Open-Label Long-Term Safety Study of Inhaled Nitric Oxide (iNO) for Pulmonary Arterial Hypertension (PAH)

DETAILED DESCRIPTION:
An open-label, long-term study to evaluate the safety of inhaled nitric oxide (iNO) in subjects with pulmonary arterial hypertension (PAH) who participated in IK-7001-PAH-201 and PULSE-PAH-004 to provide these patients with continued access to chronic iNO until the time of approval or development of iNO in PAH is discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form prior to the initiation of any study mandated procedures or assessments.
* PAH subjects who have completed all EOS assessments in IK-7001-PAH-201 and PULSE-PAH-004 and have continued drug/device usage.
* Subjects are willing and considered in the judgement of the Investigator able to use the INOpulse device continuously for up to 24 hours per day.
* All female subjects must be willing to continue to take adequate precaution to avoid pregnancy.
* Subjects in need for continued treatment with iNO in the opinion of the treating physician and agreement from Sponsor.

Exclusion Criteria:

* Subjects who require treatment with riociguat
* Subjects who early discontinued drug/device usage due to withdrawal of consent or an AE requiring termination from treatment in IK-7001-PAH-201

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Serious Adverse Events | Through Study Completion, anticipated 3 years
  Incidence of Serious Adverse Events from baseline to end of study
Incidence of INOpulse device malfunction and/or device failure leading to an AE | Through Study Completion, anticipated 3 years
  Incidence of INOpulse device malfunction and/or device failure leading to an AE from baseline to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Ashika Ahmed, MD, Study Director — Bellerophon Therapeutics
Locations (17):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - West Los Angeles VA Healthcare Center, Los Angeles, California
  - University of Colorado Denver, Aurora, Colorado
  - Cleveland Clinic Florida, Weston, Florida
  - University of Maryland Medical Center, Baltimore, Maryland
  - Mount Sinai Beth Israel, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - UC Health University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Wexner Medical Center, Columbus, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Fernando Torres, MD, Dallas, Texas
  - Intermountain Medical Center, Murray, Utah
- Canada (4):
  - Peter Lougheed Centre, Calgary, Alberta
  - University of Alberta Hospitals - MAHI, Edmonton, Alberta
  - Lawson Clinical Research Services, London, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No